CLINICAL TRIAL: NCT02993406
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Effects of Bempedoic Acid (ETC-1002) on the Occurrence of Major Cardiovascular Events in Patients With, or at High Risk for, Cardiovascular Disease Who Are Statin Intolerant
Brief Title: Evaluation of Major Cardiovascular Events in Participants With, or at High Risk for, Cardiovascular Disease Who Are Statin Intolerant Treated With Bempedoic Acid (ETC-1002) or Placebo
Acronym: CLEAR Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-043
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Statin Adverse Reaction
MeSH Terms: conditions — Cardiovascular Diseases | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bempedoic Acid 180 mg (Experimental): Bempedoic acid 180 mg tablet taken orally, once daily.
  Interventions: Drug: Bempedoic acid 180 mg tablet
- Placebo Comparator (Placebo Comparator): Matching placebo tablet taken orally, once daily
  Interventions: Drug: Matching placebo tablet

INTERVENTIONS:
Drug: Bempedoic acid 180 mg tablet — Patients take bempedoic acid 180 mg tablet orally once daily
  Other Names: ETC-1002
  Arms: Bempedoic Acid 180 mg
Drug: Matching placebo tablet — Patients take matching placebo tablet orally once daily
  Other Names: placebo comparator
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to determine if treatment with bempedoic acid (ETC-1002) versus placebo decreases the risk of cardiovascular events in participants who have or are at high risk for cardiovascular disease and are statin intolerant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* History of, or at high risk for, cardiovascular disease (CVD) including coronary artery disease, symptomatic peripheral arterial disease, cerebrovascular atherosclerotic disease, or at high risk for a cardiovascular event
* Participant-reported SI due to an adverse safety effect that started or increased during statin therapy and resolved or improved when statin therapy was discontinued resulting in an inability to tolerate:

  * 2 or more statins at any dose, or
  * 1 statin at any dose and unwilling to attempt a second statin or advised by a physician to not attempt a second statin.

Please note that participants currently tolerating very low dose statin therapy (an average daily dose of rosuvastatin <5 mg, atorvastatin <10 mg, simvastatin <10 mg, lovastatin <20 mg, pravastatin <40 mg, fluvastatin <40 mg, or pitavastatin <2 mg) are considered to be intolerant to that low dose statin. Patients may continue taking very low dose statin therapy throughout the study provided that it is stable (used for at least 4 weeks prior to screening) and well tolerated.

* Written confirmation by both participant and investigator that the participant is statin intolerant as defined above, aware of the benefit of statin use to reduce the risk of MACE including death, and also aware that many other participants who are unable to tolerate a statin are able to tolerate a different statin or dose.
* Men and nonpregnant, nonlactating women
* Fasting blood LDL-cholesterol ≥ 100 (2.6 mmol/L) at screening

Exclusion Criteria:

* Fasting blood triglycerides greater than 500 mg/dL (5.6 mmol/L) at screening
* Recent (within 90 days of screening) history of major cardiovascular events, transient ischemic attack (TIA), or unstable or symptomatic cardiac arrhythmia
* History of severe heart failure
* Uncontrolled hypertension or uncontrolled diabetes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13970 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (883):
- United States (249):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Pell City, Alabama
  - Tuscumbia, Alabama
  - Chandler, Arizona
  - Cottonwood, Arizona
  - Fountain Hills, Arizona
  - Gilbert, Arizona
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Carlsbad, California
  - Huntington Beach, California
  - Lincoln, California
  - Long Beach, California
  - Northridge, California
  - Oceanside, California
  - Rancho Cucamonga, California
  - San Diego, California
  - Santa Ana, California
  - Santa Rosa, California
  - Torrance, California
  - Vista, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Littleton, Colorado
  - Loveland, Colorado
  - Hamden, Connecticut
  - Hartford, Connecticut
  - North Haven, Connecticut
  - Stamford, Connecticut
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Clearwater, Florida
  - Crystal River, Florida
  - Fleming Island, Florida
  - Fort Lauderdale, Florida
  - Greenacres City, Florida
  - Hialeah, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Lake Worth, Florida
  - Largo, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - North Miami Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Ponte Vedra, Florida
  - Port Charlotte, Florida
  - Safety Harbor, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Covington, Georgia
  - Cumming, Georgia
  - Dunwoody, Georgia
  - Gainesville, Georgia
  - Macon, Georgia
  - Savannah, Georgia
  - Tucker, Georgia
  - Woodstock, Georgia
  - Meridian, Idaho
  - Champaign, Illinois
  - Chicago, Illinois
  - Gurnee, Illinois
  - Jerseyville, Illinois
  - Olympia Fields, Illinois
  - Rock Island, Illinois
  - Rockford, Illinois
  - Anderson, Indiana
  - Elkhart, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Munster, Indiana
  - Richmond, Indiana
  - Council Bluffs, Iowa
  - Iowa City, Iowa
  - Waterloo, Iowa
  - West Des Moines, Iowa
  - Hutchinson, Kansas
  - Kansas City, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Paducah, Kentucky
  - Eunice, Louisiana
  - Lake Charles, Louisiana
  - New Orleans, Louisiana
  - West Monroe, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Columbia, Maryland
  - Rockville, Maryland
  - Salisbury, Maryland
  - Towson, Maryland
  - Haverhill, Massachusetts
  - Hyannis, Massachusetts
  - Buckley, Michigan
  - Cadillac, Michigan
  - Caro, Michigan
  - Grand Blanc, Michigan
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Mount Clemens, Michigan
  - Petoskey, Michigan
  - Saginaw, Michigan
  - Sterling Heights, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Richfield, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Tupelo, Mississippi
  - Bridgeton, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Fremont, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Bridgeton, New Jersey
  - Bridgewater, New Jersey
  - Flemington, New Jersey
  - Haddon, New Jersey
  - Linden, New Jersey
  - Sewell, New Jersey
  - Teaneck, New Jersey
  - Albany, New York
  - Binghamton, New York
  - Bronxville, New York
  - Buffalo, New York
  - Endwell, New York
  - Jackson Heights, New York
  - Jamaica, New York
  - Manhasset, New York
  - New Windsor, New York
  - New York, New York
  - Poughkeepsie, New York
  - Saratoga Springs, New York
  - Southampton, New York
  - Asheboro, North Carolina
  - Burlington, North Carolina
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Lenoir, North Carolina
  - Mooresville, North Carolina
  - Morehead City, North Carolina
  - Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Sanford, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Marion, Ohio
  - Maumee, Ohio
  - Middleburg Heights, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Abington, Pennsylvania
  - Beaver, Pennsylvania
  - Camp Hill, Pennsylvania
  - Johnstown, Pennsylvania
  - McMurray, Pennsylvania
  - Natrona Heights, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Smithfield, Pennsylvania
  - Uniontown, Pennsylvania
  - York, Pennsylvania
  - Cumberland, Rhode Island
  - Providence, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greer, South Carolina
  - Little River, South Carolina
  - Old Point Station, South Carolina
  - Summerville, South Carolina
  - Rapid City, South Dakota
  - Fayetteville, Tennessee
  - Greeneville, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Allen, Texas
  - Amarillo, Texas
  - Seton Heart Institute, Austin, Texas
  - Dallas, Texas
  - DeSoto, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Katy, Texas
  - Kerrville, Texas
  - Lubbock, Texas
  - McKinney, Texas
  - Odessa, Texas
  - Pearland, Texas
  - Plano, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Tyler, Texas
  - Victoria, Texas
  - Farmington, Utah
  - Layton, Utah
  - Murray, Utah
  - Orem, Utah
  - Burke, Virginia
  - Charlottesville, Virginia
  - Danville, Virginia
  - Falls Church, Virginia
  - Hampton, Virginia
  - Norfolk, Virginia
  - Roanoke, Virginia
  - Suffolk, Virginia
  - Woodbridge, Virginia
  - Bellevue, Washington
  - Green Bay, Wisconsin
  - Kenosha, Wisconsin
  - La Crosse, Wisconsin
  - Madison, Wisconsin
- Argentina (38):
  - Bahía Blanca, Buenos Aires
  - Berazategui, Buenos Aires
  - Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Coronel Suárez, Buenos Aires
  - Haedo, Buenos Aires
  - La Plata, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Morón, Buenos Aires
  - San Fernando, Buenos Aires
  - San Martín, Buenos Aires
  - Vicente López, Buenos Aires
  - Zárate, Buenos Aires
  - Villa Luro, Ciudad Autonoma Buenos Aires
  - Caba, Ciudad Autonoma
  - Ciudad Autónoma de Buenos Aire, Ciudad Autonoma
  - Córdoba, Córdoba Province
  - San Vicente, Córdoba Province
  - Godoy Cruz, Mendoza Province
  - San Rafael, Mendoza Province
  - Temperley, Partido De Lomas De Zamora
  - Rosario, Santa Fe Province
  - Rosario, Sante Fe
  - San Miguel de Tucumán, Tucumán Province
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Corrientes
  - Córdoba
  - La Plata
  - Lanús
  - Morón
  - Pilar
  - Quilmes
  - Ramos Mejía
  - Rosario
  - Salta
  - San Lorenzo
  - San Miguel de Tucumán
  - Santa Fe
- Australia (31):
  - Adamstown, New South Wales
  - Camperdown, New South Wales
  - Gosford, New South Wales
  - Liverpool, New South Wales
  - Merewether, New South Wales
  - Tumbi Vmbi, New South Wales
  - Wollongong, New South Wales
  - Auchenflower, Queensland
  - Bundaberg, Queensland
  - Chermside, Queensland
  - Milton, Queensland
  - Sherwood, Queensland
  - Sippy Downs, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Ashford, South Australia
  - Fullarton, South Australia
  - Hobart, Tasmania
  - Ballarat, Victoria
  - Box Hill, Victoria
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Frankston, Victoria
  - Langwarrin, Victoria
  - Melbourne, Victoria
  - Mildura, Victoria
  - Joondalup, Western Australia
  - Murdoch, Western Australia
  - Nedlands, Western Australia
  - Perth, Western Australia
  - Subiaco, Western Australia
- Austria (6):
  - Feldkirch
  - Graz
  - Innsbruck
  - Linz
  - Vienna
  - Wiener Neustadt
- Belgium (19):
  - Aalst
  - Antwerp
  - Brasschaat
  - Bruges
  - Brussels
  - De Pinte
  - Dendermonde
  - Edegem
  - Genk
  - Ghent
  - Halen
  - Liège
  - Mechelen
  - Merksem
  - Mons
  - Tienen
  - Turnhout
  - Wetteren
  - Yvoir
- Brazil (49):
  - Fortaleza, Ceará
  - Vitória, Espírito Santo
  - Salvador, Estado de Bahia
  - Brasília, Federal District
  - Goiânia, Goiás
  - Campo Grande, Mato Grosso do Sul
  - Belo Horizonte, Minas Gerais
  - Uberlândia, Minas Gerais
  - Curitiba, Paraná
  - Belém, Pará
  - Recife, Pernambuco
  - Boa Vista, Recife
  - Natal, Rio Grande do Norte
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Santa Maria, Rio Grande do Sul
  - Caxias do Sul, Rio Grande Du Sul
  - Porto Alegre, Rio Grande Du Sul
  - Balneário Camboriú, Santa Catarina
  - Blumenau, Santa Catarina
  - São Paulo, Sau Paulo
  - Campinas, São Paulo
  - Cotia, São Paulo
  - Jaú, São Paulo
  - Marília, São Paulo
  - Paraíso, São Paulo
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - São José dos Campos, São Paulo
  - São Paulo, São Paulo
  - Tatuí, São Paulo
  - Votuporanga, São Paulo
  - Bela Vista
  - Belo Horizonte
  - Bento Gonçalves
  - Brasília
  - Curitiba
  - Goiânia
  - Joinville
  - Maceió
  - Maringá
  - Marília
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - Santa Maria
  - São José
  - São Luís
  - São Paulo
- Bulgaria (16):
  - Blagoevgrad
  - Byala
  - Dimitrovgrad
  - Haskovo
  - Pazardzhik
  - Pernik
  - Pleven
  - Plovdiv
  - Rousse
  - Sandanski
  - Sliven
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo
  - Yambol
- Canada (20):
  - Victoria, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - Brampton, Ontario
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Oakville, Ontario
  - Peterborough, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Saint-Georges, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
  - Saint-Jérôme, Quebec
  - Victoriaville, Quebec
  - Québec
- Chile (4):
  - San Bernardo
  - Santiago
  - Temuco
  - Viña del Mar
- Colombia (12):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Cali
  - Cartagena
  - Espinal
  - Ibagué
  - Manizales
  - Medellín
  - Pereira
  - San Gil
  - Zipaquirá
- Croatia (13):
  - Čakovec
  - Dubrovnik
  - Koprivnica
  - Krapinske Toplice
  - Opatija
  - Osijek
  - Rijeka
  - Slavonski Brod
  - Varaždin
  - Virovitica
  - Zabok
  - Zadar
  - Zagreb
- Czechia (24):
  - Benátky nad Jizerou
  - Beroun
  - Brandýs nad Labem
  - Brno
  - Broumov
  - Choceň
  - Chrudim
  - Frýdek-Místek
  - Havířov
  - Havlíčkův Brod
  - Hodonín
  - Hradec Králové
  - Kolín
  - Náchod
  - Olomouc
  - Ostrava
  - Pardubice
  - Prague
  - Praha 4 - Krc
  - Přerov
  - Slaný
  - Teplice
  - Trutnov
  - Uherské Hradiště
- Denmark (11):
  - Aalborg
  - Århus N
  - Ballerup Municipality
  - Copenhagen NV
  - Esbjerg
  - Glostrup Municipality
  - Hellerup
  - Holbæk
  - Nykøbing Falster
  - Vejle
  - Viborg
- Tallinn, Estonia
- Germany (39):
  - Bad Krozingen, Baden-Wurttemberg
  - Dresden, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Munich, Bavaria
  - Wallerfing, Bavaria
  - Bad Homburg, Hesse
  - Frankfurt am Main, Hesse
  - Kassel, Hesse
  - Mainz, Hesse
  - Rodgau, Hesse
  - Schwerin, Mecklenburg-Vorpommern
  - Bielefeld, North Rhine-Westphalia
  - Bochum, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Goch, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Soest, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Altenburg, Saxony
  - Böhlen, Saxony
  - Dippoldiswalde, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Markkleeberg, Saxony
  - Wermsdorf, Saxony
  - Zwenkau, Saxony
  - Bad Homburg
  - Berlin
  - Bielefeld
  - Falkensee
  - Frankfurt
  - Hamburg
  - Hanover
  - Heidelberg
  - Mainz
  - Reinfeld
- Hungary (28):
  - Orosháza, Szentetornya
  - Baja
  - Balatonfüred
  - Balatongyörök
  - Békéscsaba
  - Budapest
  - Debrecen
  - Dombóvár
  - Gyöngyös
  - Győr
  - Gyula
  - Hajdúszoboszló
  - Kalocsa
  - Kecskemét
  - Kiskunhalas
  - Miskolc
  - Mosonmagyaróvár
  - Nagykanizsa
  - Nyíregyháza
  - Orosháza
  - Pécs
  - Polgár
  - Szekszárd
  - Szentendre
  - Szentes
  - Székesfehérvár
  - Szombathely
  - Zalaegerszeg
- India (24):
  - Hyderabad, Andhra Pradesh
  - Guwahati, Assam
  - Ahmedabad, Gujarat
  - Nadiād, Gujarat
  - Surat, Gujarat
  - Vadodara, Gujarat
  - Faridabad, Haryana
  - Gurgaon, Haryana
  - Bangalore, Karnataka
  - Belagavi, Karnataka
  - Bengaluru, Karnataka
  - Hubli, Karnatak
  - Aurangabad, Maharashtra
  - Nagpur, Maharashtra
  - Nashik, Maharashtra
  - Pune, Maharashtra
  - New Delhi, National Capital Territory of Delhi
  - Jaipur, Rajasthan
  - Chennai, Tamil Nadu
  - Coimbatore, Tamil Nadu
  - Lucknow, Uttar Pradesh
  - Noida, Uttar Pradesh
  - Kolkata, West Bengal
  - Delhi
- Latvia (6):
  - Daugavpils
  - Kuldīga
  - Ogre
  - Riga
  - Tukums
  - Ventspils
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Mexico (25):
  - Tijuana, Baja California Norte
  - Chihuahua City, Chihuahua C.P.
  - Monclova, Coahuila
  - Torreón, Coahuila
  - Pachuca, Hidalgo
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Querétaro City, Querétaro
  - Culiacán, Sinaloa
  - Mazatlán, Sinaloa
  - Mérida, Yucatán
  - Aguascalientes
  - Chihuahua City
  - Cuernavaca
  - Durango
  - Guadalajara
  - Juárez
  - Mexico City
  - Monterrey
  - Pachuca
  - Puerto Vallarta
  - Querétaro
  - Tamaulipas
  - Veracruz
- Netherlands (46):
  - Alkmaar
  - Almelo
  - Almere Stad
  - Amersfoort
  - Amstelveen
  - Amsterdam
  - Apeldoorn
  - Arnhem
  - Beverwijk
  - Blaricum
  - Delft
  - Dirksland
  - Doetinchem
  - Dordrecht
  - Ede
  - Eindhoven
  - Enschede
  - Goes
  - Gorinchem
  - Gouda
  - Hardenberg
  - Harderwijk
  - Heerlen
  - Helmond
  - Hilversum
  - Hoogeveen
  - Hoogezand
  - Hoorn
  - Leeuwarden
  - Leiden
  - Leiderdorp
  - Maastricht
  - Nijmegen
  - Purmerend
  - Roosendaal
  - Rotterdam
  - Schiedam
  - Sneek
  - The Hague
  - Tiel
  - Tilburg
  - Utrecht
  - Venlo
  - Zutphen
  - Zwijndrecht
  - Zwolle
- New Zealand (10):
  - Auckland
  - Christchurch
  - Grafton
  - Hamilton
  - Hastings
  - New Plymouth
  - Papamoa
  - Rotorua
  - Tauranga
  - Wellington
- Poland (45):
  - Włocławek, Kuyavian-Pomeranian Voivodeship
  - Krakow, Lesser Poland Voivodeship
  - Tarnów, Lesser Poland Voivodeship
  - Legnica, Lower Silesian Voivodeship
  - Wroclaw, Lower Silesian Voivodeship
  - Lublin, Lubelski
  - Katowice, Silesian Voivodeship
  - Katowice, Sląskie
  - Ruda Śląska, Sląskie
  - Bialystok
  - Brzozów
  - Bydgoszcz
  - Chełm
  - Częstochowa
  - Elblag
  - Gdansk
  - Gdynia
  - Grodzisk Mazowiecki
  - Katowice
  - Kielce
  - Krakow
  - Legnica
  - Lodz
  - Lublin
  - Nałęczów
  - Nowa Sól
  - Nowy Targ
  - Oświęcim
  - Poznan
  - Puławy
  - Płock
  - Ruda Śląska
  - Rzeszów
  - Siedlce
  - Skierniewice
  - Sopot
  - Staszów
  - Szczecin
  - Tarnów
  - Tczew
  - Torun
  - Warsaw
  - Wroclaw
  - Włocławek
  - Zamość
- Romania (23):
  - Piteşti, Argeş
  - Baia Mare, Maramureş
  - Satu Mare, Satu Mare County
  - Timișoara, Timiș County
  - Alba Iulia
  - Baia Mare
  - Baloteşti
  - Brasov
  - Brăila
  - Bucharest
  - Călăraşi
  - Cluj-Napoca
  - Craiova
  - Deva
  - Galati
  - Oradea
  - Paşcani
  - Piteşti
  - Ploieşti
  - Satu Mare
  - Târgu Mureş
  - Timișoara
  - Zalău
- Russia (26):
  - Barnaul, Altayskiy Kray
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Ivanovo
  - Kazan'
  - Kemerovo
  - Kirov
  - Kirovsk
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Orenburg
  - Perm
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Sestroretsk
  - Smolensk
  - Tomsk
  - Yaroslavl
  - Yekaterinburg
- Serbia (9):
  - Belgrade
  - Kragujevac
  - Niš
  - Pančevo
  - Smederevo
  - Sremska Mitrovica
  - Užice
  - Valjevo
  - Zaječar
- Slovakia (18):
  - Bratislava, Ružinov
  - Bardejov
  - Bratislava
  - Dolný Kubín
  - Komárno
  - Košice
  - Levice
  - Lučenec
  - Ľubochňa
  - Moldava nad Bodvou
  - Nitra
  - Nové Zámky
  - Prešov
  - Rožňava
  - Svidník
  - Šahy
  - Štúrovo
  - Žilina
- South Africa (16):
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Free State
  - Centurion, Gauteng
  - Johannesburg, Gauteng
  - Kempton Park, Gauteng
  - Pretoria, Gauteng
  - Alberton, Guateng
  - Pretoria, Guateng
  - Durban, KwaZulu-Natal
  - Merebank, KwaZulu-Natal
  - Thabazimbi, Limpopo
  - Middelburg, Mpumalanga
  - Moloto South, Mpumalanga
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- Spain (8):
  - Santiago de Compostela, La Coruña
  - A Coruña
  - Almería
  - Barcelona
  - Girona
  - Madrid
  - Málaga
  - Seville
- Turkey (Türkiye) (10):
  - Adana
  - Ankara
  - Antalya
  - Edirne
  - Eskişehir
  - Istanbul
  - Izmir
  - Kocaeli
  - Mersin
  - Sivas
- Ukraine (17):
  - Brovary
  - Cherkasy
  - Chernivtsi
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Mykolaiv
  - Odesa
  - Sumy
  - Ternopil
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhia
  - Zhytomyr
- United Kingdom (35):
  - Reading, Berkshire
  - Soham, Cambridgeshire
  - Fowey, Cornwall
  - Hayle, Cornwall
  - Torpoint, Cornwall
  - Exmouth, Devon
  - Plymouth, Devon
  - Stockton-on-Tees, Durham
  - Basildon, Essex
  - London, Greater London
  - Manchester, Greater Manchester
  - East Kilbride, Lanarkshire
  - Blackpool, Lancashire
  - Chorley, Lancashire
  - Edinburgh, Lothian Region
  - Liverpool, Merseyside
  - Airdrie, North Lanarkshire
  - Hexham, Northumberland
  - Axbridge, Somerset
  - Bath, Somerset
  - Cardiff, South Glamorgan
  - Glasgow, Strathclyde
  - Chertsey, Surrey
  - Dundee, Tayside Region
  - Birmingham, West Midlands
  - Wakefield, Yorkshire and the Humber
  - Wakefield, Yorkshire
  - Blackpool
  - Chesterfield
  - Crownhill
  - Lincoln
  - Oldham
  - Royal Leamington Spa
  - Sandbach
  - Whitby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Bilen O, Ballantyne CM. Bempedoic Acid (ETC-1002): an Investigational Inhibitor of ATP Citrate Lyase. Curr Atheroscler Rep. 2016 Oct;18(10):61. doi: 10.1007/s11883-016-0611-4. PMID 27663902
- [Background] Thompson PD, MacDougall DE, Newton RS, Margulies JR, Hanselman JC, Orloff DG, McKenney JM, Ballantyne CM. Treatment with ETC-1002 alone and in combination with ezetimibe lowers LDL cholesterol in hypercholesterolemic patients with or without statin intolerance. J Clin Lipidol. 2016 May-Jun;10(3):556-67. doi: 10.1016/j.jacl.2015.12.025. Epub 2016 Jan 6. PMID 27206943
- [Background] Thompson PD, Rubino J, Janik MJ, MacDougall DE, McBride SJ, Margulies JR, Newton RS. Use of ETC-1002 to treat hypercholesterolemia in patients with statin intolerance. J Clin Lipidol. 2015 May-Jun;9(3):295-304. doi: 10.1016/j.jacl.2015.03.003. Epub 2015 Mar 19. PMID 26073387
- [Background] Nicholls S, Lincoff AM, Bays HE, Cho L, Grobbee DE, Kastelein JJ, Libby P, Moriarty PM, Plutzky J, Ray KK, Thompson PD, Sasiela W, Mason D, McCluskey J, Davey D, Wolski K, Nissen SE. Rationale and design of the CLEAR-outcomes trial: Evaluating the effect of bempedoic acid on cardiovascular events in patients with statin intolerance. Am Heart J. 2021 May;235:104-112. doi: 10.1016/j.ahj.2020.10.060. Epub 2020 Oct 24. PMID 33470195
- [Background] Nissen SE, Lincoff AM, Brennan D, Ray KK, Mason D, Kastelein JJP, Thompson PD, Libby P, Cho L, Plutzky J, Bays HE, Moriarty PM, Menon V, Grobbee DE, Louie MJ, Chen CF, Li N, Bloedon L, Robinson P, Horner M, Sasiela WJ, McCluskey J, Davey D, Fajardo-Campos P, Petrovic P, Fedacko J, Zmuda W, Lukyanov Y, Nicholls SJ; CLEAR Outcomes Investigators. Bempedoic Acid and Cardiovascular Outcomes in Statin-Intolerant Patients. N Engl J Med. 2023 Apr 13;388(15):1353-1364. doi: 10.1056/NEJMoa2215024. Epub 2023 Mar 4. PMID 36876740
- [Background] Nissen SE, Menon V, Nicholls SJ, Brennan D, Laffin L, Ridker P, Ray KK, Mason D, Kastelein JJP, Cho L, Libby P, Li N, Foody J, Louie MJ, Lincoff AM. Bempedoic Acid for Primary Prevention of Cardiovascular Events in Statin-Intolerant Patients. JAMA. 2023 Jul 11;330(2):131-140. doi: 10.1001/jama.2023.9696. PMID 37354546
- [Derived] Nicholls SJ, Ray KK, Lincoff AM, Sarnes E, Gillard KK, Bloedon L, Migliaccio-Walle K, Elsea D, Nissen SE. Cost-Effectiveness of Bempedoic Acid in High Cardiovascular Risk Patients with Statin Intolerance: An Analysis of the CLEAR Outcomes Trial. Am J Cardiovasc Drugs. 2025 Aug 20. doi: 10.1007/s40256-025-00753-w. Online ahead of print. PMID 40833562
- [Derived] Laufs U, Lincoff AM, Nicholls SJ, Li N, Bloedon L, Sasiela WJ, Powell HA, Herout PM, Thompson PD, Nissen SE. Characteristics and outcomes of patients with and without statin-associated muscle symptoms treated with bempedoic acid in the CLEAR Outcomes trial. J Clin Lipidol. 2025 Mar-Apr;19(2):337-347. doi: 10.1016/j.jacl.2024.12.014. Epub 2024 Dec 25. PMID 39939212
- [Derived] Bays HE, Bloedon L, Brennan D, Lei L, Lincoff AM, Nicholls SJ, Plutzky J, Powell HA, Nissen SE. Bempedoic Acid for Prevention of Cardiovascular Events in People With Obesity: A CLEAR Outcomes Subset Analysis. J Am Heart Assoc. 2025 Feb 18;14(4):e037898. doi: 10.1161/JAHA.124.037898. Epub 2025 Feb 8. PMID 39921511
- [Derived] Lincoff AM, Ray KK, Sasiela WJ, Haddad T, Nicholls SJ, Li N, Cho L, Mason D, Libby P, Goodman SG, Nissen SE. Comparative Cardiovascular Benefits of Bempedoic Acid and Statin Drugs. J Am Coll Cardiol. 2024 Jul 9;84(2):152-162. doi: 10.1016/j.jacc.2024.04.048. PMID 38960508
- [Derived] Ray KK, Nicholls SJ, Li N, Louie MJ, Brennan D, Lincoff AM, Nissen SE; CLEAR OUTCOMES Committees and Investigators. Efficacy and safety of bempedoic acid among patients with and without diabetes: prespecified analysis of the CLEAR Outcomes randomised trial. Lancet Diabetes Endocrinol. 2024 Jan;12(1):19-28. doi: 10.1016/S2213-8587(23)00316-9. Epub 2023 Dec 4. PMID 38061370
- [Derived] Ridker PM, Lei L, Louie MJ, Haddad T, Nicholls SJ, Lincoff AM, Libby P, Nissen SE; CLEAR Outcomes Investigators. Inflammation and Cholesterol as Predictors of Cardiovascular Events Among 13 970 Contemporary High-Risk Patients With Statin Intolerance. Circulation. 2024 Jan 2;149(1):28-35. doi: 10.1161/CIRCULATIONAHA.123.066213. Epub 2023 Nov 6. PMID 37929602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, parallel-group study that assessed the occurrence of major adverse cardiovascular event (MACE) in participants with, or at high risk for, cardiovascular disease (CVD) who were unable to tolerate statin therapy.
Pre-assignment Details: A total of 13970 participants were enrolled from over 1250 sites in 32 countries.
Groups:
- Bempedoic Acid 180 Milligrams (mg): Participants were administered with Bempedoic acid 180 mg tablet once daily orally.
- Placebo Comparator: Participants were administered with matching Placebo tablet once daily orally.
Period: Overall Study
Arm/Group | Bempedoic Acid 180 Milligrams (mg) | Placebo Comparator
Started | 6992 | 6978
Completed | 6697 | 6620
Not Completed | 295 | 358
Not completed — Withdrawal by Subject | 170 | 196
Not completed — Physician Decision | 3 | 5
Not completed — Lost to Follow-up | 12 | 13
Not completed — Unclassifiable Response | 105 | 139
Not completed — Administrative decision | 1 | 0
Not completed — Sponsor decision | 4 | 5

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat Population is defined as all randomized participants.
Groups:
- Bempedoic Acid 180 mg: Participants were administered with Bempedoic acid 180 mg tablet once daily orally.
- Total: Total of all reporting groups
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator | Total
Number analyzed (Participants) | 6992 | 6978 | 13970
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (9.0) | 65.5 (8.9) | 65.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3361 | 3379 | 6740
  Male | 3631 | 3599 | 7230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1190 | 1143 | 2333
  Not Hispanic or Latino | 5802 | 5835 | 11637
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 240 | 247 | 487
  Asian | 130 | 136 | 266
  Native Hawaiian or Other Pacific Islander | 20 | 17 | 37
  Black or African American | 156 | 172 | 328
  White | 6397 | 6335 | 12732
  More than one race | 48 | 70 | 118
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Four Component Major Adverse Cardiovascular Events (MACE)
Description: The primary efficacy end point was a four-component composite of adjudicated MACE, defined as death from cardiovascular causes, nonfatal myocardial infarction, nonfatal stroke, or coronary revascularization, as assessed in a time-to first-event analysis.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 819 | 927
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.79 to 0.96]

2. Secondary Outcome: Number of Participants With First Occurrence of Three Component MACE
Description: The first key secondary end point was a three-component MACE, defined as death from cardiovascular causes, nonfatal myocardial infarction, or nonfatal stroke.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 575 | 663
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.0058, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.76 to 0.96]

3. Secondary Outcome: Number of Participants With First Occurrence of Myocardial Infarction
Description: Number of participants with time to first occurrence of fatal and non-fatal myocardial infarction are presented.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 261 | 334
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.0016, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.66 to 0.91]

4. Secondary Outcome: Number of Participants With Time to First Occurrence of Coronary Revascularization
Description: Number of participants with time to first occurrence of coronary revascularization are presented.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 435 | 529
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.0013, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.72 to 0.92]

5. Secondary Outcome: Number of Participants With Time to First Occurrence of Stroke
Description: Number of participants with time to first occurrence of fatal and non-fatal stroke.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 135 | 158
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.1593, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.67 to 1.07]

6. Secondary Outcome: Number of Participants With Time to Cardiovascular Death
Description: Number of participants with time to cardiovascular death are presented.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 269 | 257
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.6227, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.88 to 1.24]

7. Secondary Outcome: Number of Participants With Time to All-cause Mortality
Description: All-cause mortality is death due to any cause. Number of participants with time to all-cause mortality are presented.
Time Frame: Up to 68 months
Population: Intention-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
Number analyzed (Participants) | 6992 | 6978
Participants | 434 | 420
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg vs Placebo Comparator; Test type: Superiority; p = 0.6608, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.90 to 1.18]

ADVERSE EVENTS:
Time Frame: Up to 68 months. Serious adverse events (SAEs) and non-SAEs were collected from Safety Population. The Safety Population comprises of all randomized participants who received at least 1 dose of study medication (investigational product). Deaths were endpoints and not reported as SAEs. Negatively adjudicated non- fatal MACE events were reported as SAEs.
Description: The Safety Analysis Set (SAS) included all participants in the Full Analysis Set who received at least 1 dose of study drug. Participants in the SAS were grouped according to the actual treatment received. Out of 5 participants, 2 randomized to bempedoic acid and 3 to placebo, did not receive any treatment & were not included in the SAS; 11 participants were randomized to placebo but received ≥ to 1 dose of bempedoic acid in error, and were therefore, counted in bempedoic acid group for the SAS.
Arm/Group | Bempedoic Acid 180 mg | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 437/7001 | 420/6964
Serious Adverse Events (participants affected / at risk) | 1767/7001 | 1733/6964
Other Adverse Events (participants affected / at risk) | 5805/7001 | 5490/6964
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bempedoic Acid 180 mg (N=7001) | Placebo Comparator (N=6964)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 5 (5) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 4 (4) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 11 (11) | 6 (7)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 56 (62) | 82 (84)
Angina unstable (Cardiac disorders) | 56 (58) | 53 (54)
Anginal equivalent (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 12 (12) | 6 (6)
Arrhythmia (Cardiac disorders) | 3 (3) | 3 (3)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 2 (2)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 81 (107) | 95 (111)
Atrial flutter (Cardiac disorders) | 14 (17) | 9 (10)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 7 (8) | 6 (6)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 4 (5)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 9 (10) | 5 (6)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 56 (56) | 75 (76)
Cardiac arrest (Cardiac disorders) | 3 (4) | 7 (7)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 35 (43) | 38 (46)
Cardiac failure acute (Cardiac disorders) | 19 (21) | 20 (28)
Cardiac failure chronic (Cardiac disorders) | 16 (16) | 13 (13)
Cardiac failure congestive (Cardiac disorders) | 39 (42) | 37 (45)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 4 (4) | 2 (3)
Cardiomyopathy (Cardiac disorders) | 2 (4) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 2 (2) | 3 (3)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery disease (Cardiac disorders) | 25 (26) | 33 (34)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 4 (6)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 4 (4)
Left ventricular failure (Cardiac disorders) | 4 (4) | 7 (10)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 3 (3)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 28 (28) | 35 (35)
Myocardial ischaemia (Cardiac disorders) | 7 (7) | 10 (10)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial cyst (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 6 (7) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 14 (14) | 10 (10)
Stress cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 3 (3) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 5 (5)
Ventricular tachycardia (Cardiac disorders) | 9 (15) | 14 (15)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital ectopic pancreas (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Intestinal malrotation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Trisomy 18 (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Uterine cervix canal atresia (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 2 (2) | 3 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 3 (3)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 2 (2)
Amblyopia (Eye disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (6)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Macular rupture (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (6)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 7 (7)
Abdominal wall haematoma (Gastrointestinal disorders) | 3 (3) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis noninfective (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (3)
Colitis (Gastrointestinal disorders) | 3 (3) | 5 (5)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 5 (5)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (6)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (2)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 5 (5) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 7 (7)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 (25) | 21 (24)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 6 (6)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Hiatus hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 8 (8) | 8 (8)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal angina (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 7 (7)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal strangulation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 5 (5) | 3 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 9 (9) | 5 (5)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 7 (8)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (11) | 11 (13)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach granuloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 5 (6)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (5)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Complication of device insertion (General disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 9 (9)
Diabetes mellitus (Metabolism and nutrition disorders) | 11 (11) | 16 (16)
Facial pain (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Impaired healing (General disorders) | 3 (3) | 1 (1)
Medical device site joint inflammation (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 50 (55) | 57 (60)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0)
Treatment failure (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 2 (2) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Ampulla of Vater stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 8 (8) | 8 (8)
Bile duct stone (Hepatobiliary disorders) | 6 (6) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 2 (2) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 8 (8) | 10 (11)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 3 (3)
Cholangitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 4 (4) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 38 (39) | 15 (15)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 2 (5)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 5 (5)
Heart transplant rejection (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Acute HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 19 (19) | 8 (8)
Appendicitis perforated (Infections and infestations) | 2 (2) | 2 (2)
Arthritis bacterial (Infections and infestations) | 3 (4) | 3 (3)
Arthritis infective (Infections and infestations) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Babesiosis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 6 (6)
Bronchitis viral (Infections and infestations) | 1 (1) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 84 (86) | 90 (90)
Campylobacter colitis (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac valve vegetation (Infections and infestations) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 23 (24) | 16 (18)
Cellulitis (Infections and infestations) | 11 (11) | 21 (21)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 2 (3) | 2 (2)
Chronic sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 4 (4)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Device related bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 19 (24) | 27 (35)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 3 (3)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 4 (5) | 5 (5)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 2 (2) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Gangrene (Infections and infestations) | 7 (8) | 8 (10)
Gastric ulcer helicobacter (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (11) | 7 (7)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis yersinia (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4) | 2 (2)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 1 (1)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 8 (8) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 2 (2)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 2 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 1 (1)
Listeriosis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 2 (2) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 7 (7)
Osteomyelitis acute (Infections and infestations) | 2 (2) | 1 (1)
Osteomyelitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (3)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pericarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 5 (5) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 84 (93) | 81 (92)
Pneumonia bacterial (Infections and infestations) | 5 (5) | 4 (4)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 2 (2)
Post procedural sepsis (Infections and infestations) | 0 (0) | 2 (2)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 3 (3)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 7 (7) | 5 (5)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 6 (7)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
SARS-CoV-2 sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 24 (24) | 22 (24)
Septic encephalopathy (Infections and infestations) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 5 (5) | 8 (8)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 23 (25) | 27 (28)
Syphilis (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 23 (24) | 33 (34)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 7 (8) | 7 (7)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 3 (3) | 1 (1)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24 (33) | 27 (33)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 6 (7)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 7 (7) | 9 (9)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Joint capsule rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 5 (5) | 6 (7)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Pelvic fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pharynx radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post intensive care syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 29 (30)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 8 (9)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 4 (4) | 4 (5)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 1 (1) | 0 (0)
Angiogram (Investigations) | 0 (0) | 1 (1)
Aspiration pleural cavity (Investigations) | 1 (1) | 0 (0)
Bacterial test (Investigations) | 0 (0) | 1 (1)
Biopsy lung (Investigations) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 2 (2)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 12 (13) | 11 (13)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (3) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 3 (4) | 5 (5)
Haemoglobin decreased (Investigations) | 3 (3) | 2 (2)
Influenza B virus test positive (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 2 (2)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 3 (3) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 1 (1)
Transaminases increased (Investigations) | 3 (3) | 1 (1)
Troponin increased (Investigations) | 1 (2) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 19 (21) | 15 (15)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 9 (10)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cartilage hypertrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 (13) | 15 (16)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (11)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 71 (81) | 69 (75)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 11 (17) | 6 (7)
Pancreatitis acute (Gastrointestinal disorders) | 13 (18) | 16 (20)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 10 (12) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (6)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 4 (4)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 12 (13)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 11 (11)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 5 (5)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epithelioid sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 5 (5)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (8)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oropharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ovarian endometrioid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Thyroid cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Axonal neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Basilar artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Basilar artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 7 (7)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 23 (24)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 2 (2)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 3 (3)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 5 (6) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 21 (21) | 25 (25)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (2) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Delayed ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 6 (6)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis toxic (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 3 (3)
Epilepsy (Nervous system disorders) | 5 (8) | 2 (2)
Facial paralysis (Nervous system disorders) | 2 (2) | 2 (2)
Frontotemporal dementia (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Hemiparesis (Nervous system disorders) | 2 (2) | 3 (3)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 10 (10) | 14 (14)
Lacunar infarction (Nervous system disorders) | 4 (4) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 3 (3) | 3 (3)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 4 (4)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 5 (5) | 6 (6)
Migraine (Nervous system disorders) | 3 (7) | 2 (2)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (2) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 2 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 3 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 4 (4)
Peripheral nerve lesion (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 7 (7) | 6 (6)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 21 (21)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 3 (3) | 4 (4)
Sciatica (Nervous system disorders) | 1 (1) | 3 (3)
Seizure (Nervous system disorders) | 5 (5) | 5 (6)
Spinal claudication (Nervous system disorders) | 2 (2) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (2) | 0 (0)
Spinal cord herniation (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 4 (4) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 41 (43) | 36 (36)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 3 (3) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 3 (3) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 2 (2)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device end of service (Product Issues) | 0 (0) | 4 (4)
Device failure (Product Issues) | 2 (2) | 1 (1)
Device lead damage (Product Issues) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 1 (3) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 6 (7)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (2) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (4)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 3 (3)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 8 (9) | 8 (8)
Vertigo positional (Ear and labyrinth disorders) | 4 (4) | 4 (4)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 4 (4)
Calculus urinary (Renal and urinary disorders) | 5 (5) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 18 (21) | 14 (16)
Cholecystitis acute (Hepatobiliary disorders) | 17 (18) | 19 (19)
Chronic kidney disease (Renal and urinary disorders) | 7 (7) | 3 (3)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 2 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 4 (4)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 17 (26) | 15 (17)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 7 (7) | 6 (7)
Renal hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urate nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 2 (2)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (6) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 7 (7) | 5 (5)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 18 (18) | 14 (15)
Blood loss anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 5 (5)
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vulvovaginal adhesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 35 (37) | 29 (32)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 29 (32)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (13)
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 14 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Haematuria (Renal and urinary disorders) | 8 (8) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (12)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheobronchial dyskinesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adiposis dolorosa (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 8 (10)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 2 (4) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 5 (5)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peau d'orange (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amputee (Social circumstances) | 0 (0) | 2 (2)
Cardiac assistance device user (Social circumstances) | 1 (1) | 1 (1)
Cardiac valve prosthesis user (Social circumstances) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 2 (2) | 3 (3)
Aortic aneurysm (Vascular disorders) | 13 (13) | 9 (9)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (3)
Aortic intramural haematoma (Vascular disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 0 (0) | 1 (2)
Aortic stenosis (Vascular disorders) | 13 (14) | 5 (5)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 3 (3)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 19 (20)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 (8) | 8 (9)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7) | 10 (10)
Giant cell arteritis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 8 (8) | 11 (12)
Hypertension (Vascular disorders) | 29 (29) | 26 (30)
Hypertensive crisis (Vascular disorders) | 16 (16) | 9 (12)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 3 (3) | 6 (6)
Hypotension (Vascular disorders) | 5 (6) | 11 (11)
Hypovolaemic shock (Vascular disorders) | 4 (4) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 2 (2)
Iliac artery stenosis (Vascular disorders) | 4 (4) | 4 (4)
Intermittent claudication (Vascular disorders) | 2 (5) | 3 (3)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Labile hypertension (Vascular disorders) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 2 (3)
Penetrating atherosclerotic ulcer (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 30 (43) | 25 (40)
Peripheral artery aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 3 (4) | 5 (6)
Peripheral artery stenosis (Vascular disorders) | 3 (3) | 4 (4)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 5 (5) | 7 (7)
Peripheral vascular disorder (Vascular disorders) | 3 (4) | 9 (11)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Renovascular hypertension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 2 (2)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Varicose vein (Vascular disorders) | 2 (2) | 4 (4)
Varicose vein ruptured (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bempedoic Acid 180 mg (N=7001) | Placebo Comparator (N=6964)
COVID-19 (Infections and infestations) | 731 (756) | 801 (826)
Urinary tract infection (Infections and infestations) | 539 (802) | 515 (784)
Nasopharyngitis (Infections and infestations) | 351 (424) | 389 (462)
Arthralgia (Musculoskeletal and connective tissue disorders) | 548 (675) | 554 (722)
Back pain (Musculoskeletal and connective tissue disorders) | 404 (458) | 450 (511)
Myalgia (Musculoskeletal and connective tissue disorders) | 392 (511) | 470 (599)
Hyperuricaemia (Metabolism and nutrition disorders) | 763 (868) | 393 (435)
Diabetes mellitus (Metabolism and nutrition disorders) | 458 (509) | 435 (475)
Blood uric acid increased (Investigations) | 393 (439) | 186 (201)
Headache (Nervous system disorders) | 479 (572) | 493 (574)
Hypertension (Vascular disorders) | 747 (907) | 804 (978)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02993406/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02993406/SAP_001.pdf